CLINICAL TRIAL: NCT00178126
Title: An RCT on Preventing Pressure Ulcers With Seat Cushions
Brief Title: An RCT on Preventing Pressure Ulcers With Wheelchair Seat Cushions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, David Brienza, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0403061; R01HD041490 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-04

CONDITIONS: Pressure Ulcer
Keywords: pressure ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Segmented Foam Cushion (Active Comparator): Receive seating assessment, wheelchair and seat cushion representing the standard of care in nursing homes
  Interventions: Device: Segmented Foam Wheelchair Seat Cushion
- Skin Protection Cushion (Experimental): Receive seating assessment, wheelchair and cushion meeting CMS code for Skin Protection Wheelchair Cushion
  Interventions: Device: Skin Protection Wheelchair Seat Cushion

INTERVENTIONS:
Device: Skin Protection Wheelchair Seat Cushion — Cushion receiving CMS code for Skin Protection Wheelchair Cushion
  Other Names: ROHO, Quadtro; Sunrise Medical, Jay2 Deep Contour; Invacare, Infinity
  Arms: Skin Protection Cushion
Device: Segmented Foam Wheelchair Seat Cushion — General use class wheelchair seat cushion
  Arms: Segmented Foam Cushion

SUMMARY:
The primary aim of the proposed multi-site, randomized pressure-reducing wheelchair trial (PRWC-II) is to determine the efficacy of pressure-reducing cushions in preventing sitting-acquired pressure ulcers in the elderly, nursing home population. Positive results of the proposed trial will provide the level of evidence needed to change the standard of care to include the routine evaluation of at-risk residents for seating and positioning needs and the provision of pressure-reducing cushions as a preventive measure against sitting-acquired pressure ulcers. If our hypothesis is valid, such intervention should result in a decrease in the incidence and prevalence of sitting-acquired pressure ulcers, reduced healthcare costs, and improved quality of life.

DETAILED DESCRIPTION:
Pressure ulcers (aka pressure sores, bed sores and decubitus ulcers) are a significant healthcare problem for the growing number of United States elderly long-term care (LTC) residents. Pressure ulcers (PU) diminish quality of life, exact a devastating loss of function, increase the risk of death in geriatric populations and raise healthcare costs.

Despite Federal preventive mandates for the long-term care (LTC) setting, widespread non-compliance occurs. The last three Centers for Medicare and Medicaid Services (CMS) LTC surveys showed a cumulative increase of 21% in the number of citations issued for failure to provide proper intervention to prevent or treat pressure ulcers. Costs for the management of PU in the US likely exceed $6.4 billion annually with a prevalence of approximately 28% in the LTC population.

Estimates of the number of sitting-acquired PU in the elderly, at-risk population range from 36-50%. Several studies, including our own pilot investigation, support these estimates and have suggested that the use of wheelchair cushions designed to reduce interface pressure will reduce the incidence of sitting-acquired PU. Despite this evidence, elderly wheelchair users are not routinely evaluated for seating and positioning needs as definitive studies have not been completed to justify funding for such seating interventions. Consequently, elderly Medicare beneficiaries are being denied access to medically necessary and clinically appropriate interventions and instead are most frequently provided with convoluted or segmented-foam cushions that are not designed for pressure ulcer prevention.

The primary aim of the proposed multi-site, randomized pressure-reducing wheelchair trial (PRWC-II) is to determine the efficacy of pressure-reducing cushions in preventing sitting-acquired pressure ulcers in the elderly, nursing home population. Positive results of the proposed trial will provide the level of evidence needed to change the standard of care to include the routine evaluation of at-risk residents for seating and positioning needs and the provision of pressure-reducing cushions as a preventive measure against sitting-acquired pressure ulcers. If our hypothesis is valid, such intervention should result in a decrease in the incidence and prevalence of sitting-acquired pressure ulcers, reduced healthcare costs, and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 65 and older
* use wheelchair > 6 hours per day
* no pressure ulcer on sitting surface
* Braden score of 18 or less
* combined activity and mobility Braden sub-score of 5 or less

Exclusion Criteria:

* Body Weight exceeds 250 lbs.
* Hip Width exceeds 20 inches
* does not meet all criteria of seating needs assessment
* current use of cushioning material or wheelchair better than study devices

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 232 (Actual)
Dates: Start 2004-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Brienza, Ph.D., Principal Investigator — University of Pittsburgh; Sheryl Kelsey, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brienza D, Kelsey S, Karg P, Allegretti A, Olson M, Schmeler M, Zanca J, Geyer MJ, Kusturiss M, Holm M. A randomized clinical trial on preventing pressure ulcers with wheelchair seat cushions. J Am Geriatr Soc. 2010 Dec;58(12):2308-14. doi: 10.1111/j.1532-5415.2010.03168.x. Epub 2010 Nov 10. PMID 21070197

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Segmented Foam Cushion | Skin Protection Cushion
Started | 119 | 113
Completed | 94 | 86
Not Completed | 25 | 27
Not completed — Lost to Follow-up | 21 | 21
Not completed — did not receive intervention | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Segmented Foam Cushion | Skin Protection Cushion | Total
Number analyzed (Participants) | 119 | 113 | 232
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 119 | 113 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 86.5 (7.7) | 86.7 (7.4) | 86.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 91 | 197
  Male | 13 | 22 | 35
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.0 (5.2) | 24.6 (4.4) | 24.8 (4.8)
Incontinence [Number; unit: participants] | 97 | 97 | 194

OUTCOME MEASURES:

1. Primary Outcome: Sitting-induced Pressure Ulcers
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Segmented Foam Cushion | Skin Protection Cushion
Number analyzed (Participants) | 119 | 113
participants | 8 | 1
Statistical Analysis 1: Comparison: Segmented Foam Cushion vs Skin Protection Cushion; Test type: Superiority or Other; p = 0.04, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Segmented Foam Cushion | Skin Protection Cushion
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/113
Other Adverse Events (participants affected / at risk) | 0/119 | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No